CLINICAL TRIAL: NCT00669123
Title: Fase IV Clinical Trial to Evaluate Chondroitin Sulphate Efficacy and Safety in Patients With Knee Osteoarthritis and Psoriasis
Brief Title: Chondroitin Sulphate Efficay/Safety in Patients With Knee Osteoarthritis and Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Dr Josep Vergés Milano, Scientific Medical Director, Bioiberica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS/IV/PSO/ART
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis; Psoriasis; Joint Diseases; Muskuloskeletal Diseases; Skin Diseases
Keywords: Chondroitin sulphate; Knee osteoarthritis; Psoriasis
MeSH Terms: conditions — Osteoarthritis; Psoriasis; Joint Diseases; Skin Diseases; Osteoarthritis, Knee | interventions — Chondroitin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental): Chondroitin sulphate
  Interventions: Drug: Chondroitin sulphate

INTERVENTIONS:
Drug: Chondroitin sulphate — Chondroitin sulphate 800 mg/day
  Other Names: Condrosan
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpouse of this study is to determine the efficacy and safety of chondroitin sulphate conventional treatment in patients with both knee osteoarthritis and plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee OA according to ACR criteria;
* OA of radiological stages 1 to 3 according to Kellgren-Lawrence;
* VAS of pain ≥30;
* PASI ≥ 5.

Exclusion Criteria:

* Known allergy to chondroitin sulphate;
* Other bone and articular diseases such as chondrocalcinosis, Paget's disease, rheumatoid arthritis, psoriatic arthritis, acromegaly, hemochromatosis, Wilson's disease;
* Patients with skin conditions that could interfere in the clinical trial evaluation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)

PRIMARY OUTCOMES:
Huskisson Visual Analogue Scale | Monthly
Psoriasis Area and Severity Index | Monthly

SECONDARY OUTCOMES:
Lequesne Index | Monthly
Use of rescue medication | Monthly
SF-36 Health Questionaire | 3 months
Overall Lession Severity Scale | Monthly
Physician's Global Assessment of improvement | Monthly
Histological assessment of skin biopsies | 3 months
Dermatology Life Quality Index | Monthly
Tolerability | Monthly
Adverse events | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Pere Benito, MD, Principal Investigator — Hospital del Mar; Montserrat Pérez, MD, Principal Investigator — Instituto Poal de Reumatología; Ingrid Möller, MD, Principal Investigator — Instituto Poal de Reumatología
Locations (2):
- Spain (2):
  - Hospital del Mar, Barcelona, Barcelona
  - Instituto Poal de Reumatología, Barcelona, Barcelona

REFERENCES:
- [Derived] Moller I, Perez M, Monfort J, Benito P, Cuevas J, Perna C, Domenech G, Herrero M, Montell E, Verges J. Effectiveness of chondroitin sulphate in patients with concomitant knee osteoarthritis and psoriasis: a randomized, double-blind, placebo-controlled study. Osteoarthritis Cartilage. 2010 Jun;18 Suppl 1:S32-40. doi: 10.1016/j.joca.2010.01.018. Epub 2010 May 10. PMID 20399899